CLINICAL TRIAL: NCT04108208
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase IV Study of Apalutamide in Chinese Participants With Non-Metastatic Castration-Resistant Prostate Cancer (NM-CRPC)
Brief Title: A Study of Apalutamide in Chinese Participants With Non Metastatic Castration Resistant Prostate Cancer (NM-CRPC)
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR108660; 56021927PCR4007 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Results first posted 2025-03-28 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; Androgen Antagonists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apalutamide 240 milligram (mg) plus ADT (Experimental): Participants will receive apalutamide 240 mg orally daily from Day 1 of Cycle 1 until disease progression, unacceptable toxicity, withdrawal of consent, death or termination of the study along with androgen-deprivation therapy (ADT). Each treatment cycle will consist of 28 days.
  Interventions: Drug: Apalutamide; Drug: Androgen-deprivation Therapy (ADT)
- Placebo plus ADT (Placebo Comparator): Participants will receive matching placebo daily along with ADT from Cycle 1 Day 1 until disease progression, unacceptable toxicity, withdrawal of consent, death or termination of the study. Participants who do not have distant metastasis will switch to treatment with apalutamide after completion of 5 cycles of placebo treatment. Participants who have prostate-specific antigen (PSA) progression prior to completion of 5 cycles of study treatment, will cross over to apalutamide at the time of PSA progression. Each treatment cycle will consist of 28 days.
  Interventions: Drug: Placebo; Drug: Androgen-deprivation Therapy (ADT)

INTERVENTIONS:
Drug: Apalutamide — Apalutamide 240 mg (4*60 mg tablets) will be administrated orally once daily.
  Other Names: JNJ-56021927; ARN-509
  Arms: Apalutamide 240 milligram (mg) plus ADT
Drug: Placebo — Matching placebo will be administered orally.
  Arms: Placebo plus ADT
Drug: Androgen-deprivation Therapy (ADT) — Participants will continue to receive ADT with gonadotrophin-releasing hormone agonists (GnRHa) who have not been surgically castrated.

SUMMARY:
The purpose of this study is to compare the improvement in time to prostate specific antigen (PSA) progression (TTPP, as defined by Prostate Cancer Working Group 2 [PCWG2]) of apalutamide versus placebo in Chinese participants with high-risk non-metastatic castration resistant prostate cancer (NM-CRPC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features, with high risk for development of metastases, defined as prostate-specific antigen doubling time (PSADT) less than or equals to (<=) 10 months. PSADT is calculated using at least 3 prostate-specific antigen (PSA) values obtained during continuous androgen deprivation therapy (ADT)
* Castration-resistant prostate cancer (PC) demonstrated during continuous ADT, defined as 3 PSA rises at least 1 week apart, with the last PSA greater than (>) 2 nanogram per milliliter (ng/mL)
* Surgically or medically castrated, with testosterone levels of less than (<) 50 nanogram per deciliter (ng/dL). If the participant is medically castrated, continuous dosing with gonadotropin releasing hormone analog (GnRHa) must have been initiated at least 4 weeks prior to randomization and must be continued throughout the study to maintain castrate levels of testosterone
* Participants who received a first-generation anti-androgen (example: bicalutamide, flutamide, nilutamide) must have at least a 4-week washout prior to randomization and must show continuing disease progression (an increase in PSA) after washout
* At least 4 weeks must have elapsed from major surgery or radiation therapy prior to randomization

Exclusion Criteria:

* Presence of distant metastases, including central nervous system (CNS) and vertebral or meningeal involvement, or history of distant metastases. Exception: Pelvic lymph nodes <2 centimeter in short axis (N1) located below the iliac bifurcation are allowed
* Symptomatic loco-regional disease requiring medical intervention, such as moderate or severe urinary obstruction or hydronephrosis, due to primary tumor (example, tumor obstruction of bladder trigone)
* Prior treatment with cytochrome P450 17 alpha-hydroxylase/17,20-lyase (CYP17) inhibitors (example: abiraterone acetate, orteronel, galerterone, ketoconazole, aminoglutethimide) for PC
* Prior chemotherapy for PC, except if administered in the adjuvant/neoadjuvant setting
* Prior treatment with second generation anti-androgens (example, enzalutamide)
* History of seizure or condition that may pre-dispose to seizure (example: prior stroke within 1 year prior to randomization, brain arteriovenous malformation, schwannoma, meningioma, or other benign CNS or meningeal disease which may require treatment with surgery or radiation therapy)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2026-06-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (27):
- China (27):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Beijing Friendship Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Beijing Hospital, Beijing
  - Hunan Cancer hospital, Changsha
  - Sichuan Provincial Peoples Hospital, Chengdu
  - Chongqing University Cancer Hospital, Chongqing
  - Fujian Medical University Union Hospital, Fuzhou
  - Sun Yat-Sen Memorial Hospital Sun Yat-sen University, Guangzhou
  - Guangzhou First Municipal People's Hospital, Guangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - The First Affiliated Hospital Zhejiang University College of Medicine, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Nanjing Drum Tower Hospital, Nanjing
  - The First Affiliated Hospital of Ningbo University, Ningbo
  - Cancer Hospital, FuDan University, Shanghai
  - Shanghai Zhongshan Hospital, Shanghai
  - Huashan Hospital Fudan University, Shanghai
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - The Fifth People's Hospital of Shanghai, Fudan University, Shanghai
  - Huadong Hospital Affiliated to Fudan University, Shanghai
  - First Affiliated Hospital SooChow University, Suzhou
  - TongJi Hospital of TongJi Medical College of Huazhong University of Science & Technology, Wuhan
  - Wuxi People s Hospital, Wuxi
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Results are currently reported till primary completion date (01 Jun 2023). Post completing end of treatment (EoT, 30 days after last dose of study treatment) visit, participants entered post-treatment followup phase and remained in study until death, recording of development of symptomatic progression, initiation of any new systemic anticancer therapies, withdrawal of consent or study termination. Follow-up phase is still ongoing and thus remaining results will be posted upon study completion.
Groups:
- Placebo Plus Androgen-deprivation Therapy (ADT): Participants received placebo matching to apalutamide tablets orally once daily along with ADT of Cycle 1 Day 1 until disease progression, unacceptable toxicity, withdrawal of consent, death or termination of the study. Each treatment cycle was of 28 days. Participants who did not have distant metastasis were switched to receive apalutamide + ADT from Cycle 6 Day 1 and those who had prostate-specific antigen (PSA) prior to completion of first 5 cycles crossed over to receive apalutamide + ADT at the time of PSA progression. Treatment continued until disease progression, unacceptable toxicity, withdrawal of consent, death or termination of the study by the sponsor.
- Apalutamide 240 mg Plus ADT: Participants received apalutamide 240 milligrams (mg) tablets (4 tablets of 60 mg) orally once daily along with ADT from Cycle 1 Day 1 until disease progression, unacceptable toxicity, withdrawal of consent, death or termination of the study. Each treatment cycle was of 28 days.
Period: Overall Study
Arm/Group | Placebo Plus Androgen-deprivation Therapy (ADT) | Apalutamide 240 mg Plus ADT
Started | 25 | 50
Crossed-over to Apalutamide | 22 | 0
Completed | 0 | 0
Not Completed | 25 | 50
Not completed — Withdrawal by Subject | 2 | 6
Not completed — other-ongoing | 20 | 40
Not completed — Death | 1 | 4
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Plus Androgen-deprivation Therapy (ADT) | Apalutamide 240 mg Plus ADT | Total
Number analyzed (Participants) | 25 | 50 | 75
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74.5 (7.82) | 75.1 (7.90) | 74.9 (7.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 25 | 50 | 75
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 25 | 50 | 75
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 25 | 50 | 75

OUTCOME MEASURES:

1. Primary Outcome: Time to Prostate Specific Antigen (PSA) Progression (TTPP) Based on Prostate Cancer Working Group 2 (PCWG2) Criteria
Description: Time to prostate specific antigen progression (TTPP) was defined as the time from randomization to the first date of documented PSA progression based on PCWG2 criteria. PCWG2 was defined as the PSA progression as 1) the date that a 25 percent (%) or greater increase and an absolute increase of 2 nanograms per milliliter (ng/mL) or more from the Nadir was documented, which was confirmed by a second value obtained 3 or more weeks later. 2) Where no decline from baseline was documented as a 25% increase from the baseline value along with an increase in absolute value of 2 ng/mL or more after 12 week of treatment. Kaplan-Meier method was used for the analysis.
Time Frame: From randomization until first documented PSA progression (up to 3 years 3 months)
Population: The Intent-to-Treat (ITT) analysis set included all randomized participants and were classified according to their assigned treatment group, regardless of the actual treatment received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo Plus Androgen-deprivation Therapy (ADT) | Apalutamide 240 mg Plus ADT
Number analyzed (Participants) | 25 | 50
Months | NA [3.55 to NA] — Here, "NA" denotes in the median and upper limit of 95% confidence interval (CI) were not estimable due to insufficient number of participants with events. | NA [25.76 to NA] — Here, "NA" denotes in the median and upper limit of 95% CI were not estimable due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Placebo Plus Androgen-deprivation Therapy (ADT) vs Apalutamide 240 mg Plus ADT; Test type: Superiority; p = 0.0052, Log Rank; Hazard Ratio (HR) = 0.233, 95% CI 2-sided [0.077 to 0.705]

2. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Time Frame: Up to 6 years 4 months
Reporting Status: Not Posted, anticipated posting 2027-06

3. Secondary Outcome: Number of Participants With Grade 3 or Higher Abnormalities in Laboratory Values
Time Frame: Up to 6 years 4 months
Reporting Status: Not Posted, anticipated posting 2027-06

4. Secondary Outcome: Percentage of Participants Who Achieved Prostate Specific Antigen (PSA) Response (>=50% PSA Reduction)
Time Frame: Up to 6 years 4 months
Reporting Status: Not Posted, anticipated posting 2027-06

5. Secondary Outcome: Plasma Concentration of Apalutamide and Its Metabolite (N-desmethyl Apalutamide)
Time Frame: Presdose: Day 1 of Cycles 1, 2, 3, and 6; 2 hours postdose: Day 1 of Cycles 1 and 3
Reporting Status: Not Posted, anticipated posting 2027-06

ADVERSE EVENTS:
Time Frame: Serious adverse events (AEs) and other AEs: From Cycle 1 Day 1 up to 30 days post last dose of study drug (up to 38.3 months); all-cause mortality: from Cycle 1 Day 1 up to 3 years and 3 months
Description: The safety analysis set included all randomized participants who had received at least 1 dose of study drug, with treatment assignments designated according to actual study treatment received. "All participants: Apalutamide" 240 mg Plus ADT arm presents combined data for participants treated with Apalutamide + ADT which included participants from original apalutamide arm and those who crossed over from placebo arm.
Groups:
- Placebo + ADT to Apalutamide + ADT: In placebo arm, participants who did not have distant metastasis after completion of 5 cycles of placebo plus ADT treatment and participants who had PSA progression prior to completion of 5 cycles of study treatment were crossed over to apalutamide 240 mg + ADT treatment and were treated until disease progression, unacceptable toxicity, withdrawal of consent, death or termination of the study.
- All Participants: Apalutamide 240 mg Plus ADT: All participants who received apalutamide 240 mg in arm 'Apalutamide 240 mg Plus ADT' and arm 'Placebo + ADT to Apalutamide + ADT".
Arm/Group | Placebo Plus Androgen-deprivation Therapy (ADT) | Apalutamide 240 mg Plus ADT | Placebo + ADT to Apalutamide + ADT | All Participants: Apalutamide 240 mg Plus ADT
All-Cause Mortality (participants affected / at risk) | 1/25 | 4/50 | 0/22 | 4/72
Serious Adverse Events (participants affected / at risk) | 4/25 | 20/50 | 5/22 | 25/72
Other Adverse Events (participants affected / at risk) | 11/25 | 47/50 | 21/22 | 68/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Plus Androgen-deprivation Therapy (ADT) (N=25) | Apalutamide 240 mg Plus ADT (N=50) | Placebo + ADT to Apalutamide + ADT (N=22) | All Participants: Apalutamide 240 mg Plus ADT (N=72)
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Atrioventricular Block Complete (Cardiac disorders) | 0 | 1 | 0 | 1
Mixed Deafness (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Gastritis Erosive (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 1
Covid-19 (Infections and infestations) | 0 | 2 | 1 | 3
Pneumonia (Infections and infestations) | 0 | 5 | 0 | 5
Sepsis (Infections and infestations) | 0 | 0 | 1 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Osteoporotic Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Gastrointestinal Stromal Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Cerebral Infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Hypoxic-Ischaemic Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 1
Suicide Attempt (Psychiatric disorders) | 1 | 0 | 0 | 0
Calculus Bladder (Renal and urinary disorders) | 0 | 2 | 0 | 2
Angiolymphoid Hyperplasia with Eosinophilia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Dermatitis Exfoliative Generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Plus Androgen-deprivation Therapy (ADT) (N=25) | Apalutamide 240 mg Plus ADT (N=50) | Placebo + ADT to Apalutamide + ADT (N=22) | All Participants: Apalutamide 240 mg Plus ADT (N=72)
Anaemia (Blood and lymphatic system disorders) | 3 | 15 | 5 | 20
Leukopenia (Blood and lymphatic system disorders) | 0 | 9 | 3 | 12
Lymphopenia (Blood and lymphatic system disorders) | 1 | 4 | 1 | 5
Neutropenia (Blood and lymphatic system disorders) | 0 | 4 | 2 | 6
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 0 | 3
Toothache (Gastrointestinal disorders) | 0 | 2 | 2 | 4
Fatigue (General disorders) | 0 | 3 | 1 | 4
Malaise (General disorders) | 0 | 4 | 0 | 4
Oedema Peripheral (General disorders) | 0 | 3 | 0 | 3
Pyrexia (General disorders) | 1 | 0 | 4 | 4
Covid-19 (Infections and infestations) | 0 | 6 | 5 | 11
Pneumonia (Infections and infestations) | 1 | 4 | 0 | 4
Suspected Covid-19 (Infections and infestations) | 0 | 0 | 2 | 2
Fracture (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 3
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 5 | 2 | 7
Alanine Aminotransferase Increased (Investigations) | 1 | 3 | 1 | 4
Aspartate Aminotransferase Increased (Investigations) | 2 | 2 | 1 | 3
Blood Thyroid Stimulating Hormone Increased (Investigations) | 0 | 3 | 0 | 3
Low Density Lipoprotein Increased (Investigations) | 0 | 3 | 0 | 3
Weight Decreased (Investigations) | 0 | 10 | 2 | 12
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 4 | 1 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 10 | 3 | 13
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 5 | 0 | 5
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 3 | 1 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3 | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 3
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 4
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 3
Eczema (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 5 | 1 | 6
Rash (Skin and subcutaneous tissue disorders) | 3 | 14 | 4 | 18
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 3
Hypertension (Vascular disorders) | 2 | 11 | 3 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2022-06-20): https://cdn.clinicaltrials.gov/large-docs/08/NCT04108208/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-12): https://cdn.clinicaltrials.gov/large-docs/08/NCT04108208/SAP_001.pdf